CLINICAL TRIAL: NCT00010413
Title: Phase II Study of High-Dose Cyclophosphamide in Patients With Refractory Pemphigus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15674; JHOC-J9912; JHOC-99022610
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-10

CONDITIONS: Pemphigus
Keywords: immunologic disorders and infectious disorders; pemphigus; rare disease
MeSH Terms: conditions — Pemphigus; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Cyclophosphamide; Filgrastim

INTERVENTIONS:
Drug: cyclophosphamide
Drug: filgrastim

SUMMARY:
OBJECTIVES:

I. Determine the response rate and 1-year event-free survival of patients with refractory pemphigus treated with high-dose cyclophosphamide.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive cyclophosphamide IV on days 1-4 and filgrastim (G-CSF) beginning on day 10 and continuing until blood counts recover.

Patients are followed monthly for 6 months, every 2 months for 6 months, every 4 months for a year, and then annually thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Definitive diagnosis of pemphigus, including all of the following: Typical clinical lesions Histologically proven by skin or mucous membrane biopsy Pemphigus IgG autoantibodies in skin or mucous membrane by direct immunofluorescence (IF) Circulating pemphigus IgG autoantibodies in serum by indirect IF

Dependence on high-dose corticosteroids

Persistent disease activity despite treatment with mycophenolate mofetil or azathioprine, or inability to tolerate these drugs (for paraneoplastic pemphigus, persistent disease activity despite treatment with cyclosporine)

--Prior/Concurrent Therapy--

No concurrent cytotoxic therapy

--Patient Characteristics--

Performance status: Karnofsky 20-100%

Renal: Creatinine no greater than 2.5 mg/dL

Cardiovascular: LVEF at least 40%

Pulmonary: FVC, FEV1, or DLCO at least 50% predicted

Other: Not pregnant Fertile patients must use effective contraception during and for 9 months after study Not preterminal or moribund

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 1999-04; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant J. Anhalt, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States